CLINICAL TRIAL: NCT03501524
Title: Video_ Assisted Thoracoscopic Surgery Evacuation Compared to Reinsertion of Thoracostomy Tube in Persistent Traumatic Haemothorax
Brief Title: VATS Evacuation Compared to Reinsertion of Thoracostomy Tube in Persistent Traumatic Haemothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Emad El-Dein Omar, resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17100227
Record Dates: First submitted 2018-04-08; First posted 2018-04-18 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Hemothorax; Traumatic
MeSH Terms: conditions — Hemothorax

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VATS evacuation (Experimental): patients selected for VATS after failure of first thoracostomy tube drainage
  Interventions: Device: VATS evacuation; Device: thoracostomy tube
- thoracostomy tube (Experimental): patients selected for thoracostomy tube reinsertion after failure of drainage with first thoracostomy tube
  Interventions: Device: VATS evacuation; Device: thoracostomy tube

INTERVENTIONS:
Device: VATS evacuation — the patient will be randomized to a Video-Assisted thoracoscopy for retained haemothorax
Device: thoracostomy tube — the patient is randomized to reinsertion of a Thoracostomy Tube for retained haemothorax
  Other Names: intercostal tube reinsertion

SUMMARY:
This is prospective, randomized study comparing VATS (video- Assisted Thoracoscopy) to reinsertion of a thoracostomy tube in patients with persistent traumatic haemothorax. The incidence varies and can be as high as 20%, but in most studies is found to be 1-4% after initial tube thoracostomy for chest trauma. The most accepted complication of retained hemothorax is empyema.Retained hemothorax treatment started by physiotherapy and early withdrawal of tube thoracostomy which lead to more complications as empyema, fibro thorax/entrapped lung, flail chest and diaphragmatic hernia. Early VATS is an alternative treatment for retained hemothorax with evidence that it is a superior intervention when compared to a second tube thoracostomy.

DETAILED DESCRIPTION:
Traumatic injuries are a significant cause of morbidity and mortality in our society.At Assiut university hospitals, chest injuries (17.7%) considered as second cause of mortality after head injuries (34.6%) of registered deaths by cause of injury at trauma unit, Assiut university hospitals in a study conducted between,2002-2009. In United States, thoracic injuries are the primary factor in approximately 35% of these deaths, one -third of which occur immediately following the injury, and are contributing in nearly 75% of trauma -related deaths. Up to 15% of patients who sustain thoracic trauma undergo emergent thoracotomy for resuscitation, massive hemothorax, cardiac tamponade, large thoracic wounds, major thoracic vascular injuries, tracheobronchial injuries, or evidence of esophageal injury. The remaining 85-90% of patients who reach the emergency department does not require emergent thoracotomy are initially managed with tube thoracostomy, pain control, pulmonary toilet, and observation .Patients failing this management ultimately require elective thoracotomy for further evaluation and treatment(clotted hemothorax, empyema and diaphragmatic hernia. The current role of VATS in trauma includes evaluation and control of continued chest tube bleeding, early evacuation of retained hemothorax, evacuation and decortication of posttraumatic empyemas, evaluation and limited treatment of suspected diaphragm injuries, evaluation and treatment of persistent air leaks, and evaluation of mediastinal injuries.

ELIGIBILITY:
Inclusion Criteria:

We include for the study all patients admitted to Assiut university hospitals during the time of the study that proved persistent haemothorax that with criteria:

1. Ages that are eligible for study are between 18years to 60 years (adult)
2. Both genders will be included to study.
3. Clinical and radiological diagnosis of persistent haemothorax.
4. Thoracostomy tube blockage or failure to drain within 5-7days.

Exclusion Criteria:

1. More than one thoracostomy tube drainage in the same attempt side.
2. Unable to consent to trial.
3. Coexisting pathology requiring other interventions.
4. Patients that need urgent interventions (hemodynamically unstable, empyema and flail chest).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalization | average 5-7 days
  number of days spent

SECONDARY OUTCOMES:
number of patients developed empyema | through one month
  the study will be monitored for septic complications , specially empyema.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Khalil salama Ayyad, PHD, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt